CLINICAL TRIAL: NCT00403585
Title: A Phase IV, Open Label, Single Arm, Multicenter, Extension Study of Adefovir Dipivoxil for Korean Patients With Chronic Hepatitis B(CHB) Who Have Completed ADF 103814
Brief Title: Study of Adefovir Dipivoxil for Korean Patients With Chronic Hepatitis B(CHB) Who Have Completed ADF 103814
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADF108005; update with ADF103814
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Results first posted 2010-11-24 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-11

CONDITIONS: Hepatitis B, Chronic; Chronic Hepatitis B
Keywords: Adefovir Dipivoxil(Hepsera); Chronic Hepatitis B (CHB)
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adefovir dipivoxil 10mg

SUMMARY:
This is an open label, single-arm, multi-centre extension study for Korean patients with chronic hepatitis B and compensated liver disease who have completed one-year adefovir dipivoxil treatment in ADF103814. The objective is to assess clinical efficacy and safety of long term (up to 3 years) adefovir dipivoxil 10mg therapy.

ELIGIBILITY:
Inclusion Criteria:

Subject has completed ADF103814 and continues with adefovir dipivoxil treatment via prescription without interruption prior enrolment in this extension study.

Availability and willingness of subject to provide written informed consent.

Exclusion Criteria:

Use of immunosuppressive therapy requiring use of more than 5mg of prednisolone(or equivalent) per day, immunomodulatory therapy (including interferon or thymosin) or systemic cytotoxic agents during the study.

Previous or current lamivudine or antiviral therapy Clinical signs of decompensated liver disease as indicated by the protocol Inadequate haematological function defined by the protocol - Documented evidence of active liver disease due to other causes Hepatocellular carcinoma as evidenced by the protocol Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. This would include any uncontrolled clinically significant renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders or cancer.

Active alcohol or drug abuse or history of alcohol or drug abuse considered by the investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.

Planned for liver transplantation Therapy with nephrotoxic drugs or competitors of renal excretion can be expected during the course of the study.

History of hypersensitivity to nucleoside and/or nucleotide analogues. Inability to comply with study requirements as determined by the study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., Ph.D, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study ADF108005 (NCT00403585; 80 subjects enrolled) is an extension of Study ADF103814 (104 subjects enrolled). For several outcome measures, baseline is defined as the first day of Study 103814; thus, baseline data for 104 subjects are provided, even though 80 subjects were enrolled in Study 108005.
Groups:
- Adefovir Dipivoxil: Adefovir Dipivoxil 10 mg tablets once daily
Period: Initial Treatment Phase
Arm/Group | Adefovir Dipivoxil
Started | 104
Completed | 102
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Open-Label Phase; Extension Study
Arm/Group | Adefovir Dipivoxil
Started | 80 (80 of 102 participants completing Study 103814 enrolled in extension (22 didn't continue medication))
Completed | 74
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — HBV DNA Mutation Positive | 4

BASELINE CHARACTERISTICS:
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 35.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 83
Race/Ethnicity, Customized [Number; unit: Participants] | 104

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis B Virus (HBV) DNA (log10 Copies/mL) Change From Baseline at Week 156 of Adefovir Therapy
Description: HBV DNA was tested with Roche Cobas Amplicor HBV monitor test, Lower Limit of Detection 300 copies/mL) after 3 years (156 weeks: Weeks 1-52 in Study ADF103814; Weeks 53-156 in Study 108005) of adefovir therapy). Change from baseline was calculated as the Week 156 value minus the Baseline value. Baseline is defined as the first day of study ADF103814, of which Study 108005 is an extension.
Time Frame: Baseline, Week 156
Population: Study ADF103814 Intent-to-Treat (ITT) Population: All subjects regardless of whether or not the subject completed the planned duration of the study will be analyzed with no data exclusion. As baseline is defined as the first day of study ADF103814, all 104 subjects enrolled in this study were analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 104
log10 copies/mL
  Baseline, n=104 | 7.94 (1.66)
  Week 156, n=74 | 3.89 (1.59)
  Change from Baseline | -4.16 (1.79)
Statistical Analysis 1: Comparison: Adefovir Dipivoxil; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank — The p value represents the comparison between baseline data and data at Week 156

2. Secondary Outcome: Number of Participants Achieving ALT Normalization at Week 104 & 156
Description: Alanine aminotransferase (ALT) normalization is defined as a value <= upper limit of normal (ULN) range based on the set of subjects with ALT>ULN at baseline. The normal range for ALT is 0-40 Units/Liter.
Time Frame: Week 104, Week 156
Population: ITT Population: some participants were not tested at Weeks 104 or 156.
Measure: Number; unit: Participants
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 77
Participants
  Week 104, n=77 | 63
  Week 156, n=73 | 65

3. Secondary Outcome: Number of Participants Achieving Virological Response at Week 104 & 156
Description: Virological response is defined as HBV DNA level<300 copies/ml
Time Frame: Week 104, Week 156
Population: ITT Population: some participants were not tested at Weeks 104 or 156.
Measure: Number; unit: Participants
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 77
Participants
  Week 104, n=77 | 20
  Week 156, n=73 | 24

4. Secondary Outcome: HBV DNA Levels at Each Collection Time Point From Baseline Through Week 156
Description: Serum HBV DNA. Baseline is defined as the first day of study ADF103814, of which Study 108005 is an extension.
Time Frame: Baseline, Weeks 68, 80, 92, 104, 120, 132, 144, 156
Population: Study ADF103814 ITT Population. As baseline is defined as the first day of study ADF103814, all 104 subjects enrolled in this study were analyzed. Some participants were not tested at various weeks.
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 104
log 10 copies/mL
  Baseline, n=104 | 7.94 (1.66)
  Week 68, n=74 | 3.90 (1.37)
  Week 80, n=73 | 3.79 (1.36)
  Week 92, n=77 | 3.99 (1.49)
  Week 104, n=76 | 3.97 (1.44)
  Week 120, n=76 | 3.88 (1.44)
  Week 132, n=78 | 3.93 (1.51)
  Week 144, n=74 | 3.97 (1.55)
  Week 156, n=73 | 3.89 (1.59)

5. Secondary Outcome: Number of Participants With HBeAg Loss, HBeAg Seroconversion, HBsAg Loss and HBsAg Seroconversion at Week 104 & 156
Description: Hepatitis B e antigen (HBeAg) loss, HBeAg seroconversion (defined as HBeAg negative and hepatitis B e antibody [HBeAb] positive), hepatitis B surface antigen (HBsAg) loss and HBsAg seroconversion (defined as HBsAg negative and hepatitis B surface antibody [HBsAb] positive). HBeAg and HBsAg seroconversion are defined as the loss (becoming negative) of HBeAg and the concurrent appearance of antibodies against HBeAg and the loss of HBsAg and the concurrent appearance of antibodies against HBsAg, respectively.
Time Frame: Week 104 and 156
Population: All participants achieving viological response, defined as an HBV DNA level ≤ 300. Some participants were not tested at various weeks.
Measure: Number; unit: Participants
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 77
Participants
  Week 104 HBeAg loss, n=77 | 23
  Week 104 HBeAg seroconversion, n=77 | 6
  Week 104 HBsAg loss, n=77 | 0
  Week 104 HBsAg seroconversion, n=77 | 0
  Week 156 HBeAg loss, n=73 | 27
  Week 156 HBeAg seroconversion, n=73 | 12
  Week 156 HBsAg loss, n=73 | 1
  Week 156 HBsAg seroconversion, n=73 | 0

6. Secondary Outcome: Safety Assessment: Number of Participants With a Serious Adverse Event and an Adverse Event
Description: The number of participants with a serious adverse event and an adverse event is reported. Refer to the adverse event section for details.
Time Frame: Treatment Phase (Weeks 53-156)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Adefovir Dipivoxil
Number analyzed (Participants) | 80
participants
  Serious adverse event | 2
  Adverse event | 43

ADVERSE EVENTS:
Arm/Group | Adefovir Dipivoxil
Serious Adverse Events (participants affected / at risk) | 2/80
Other Adverse Events (participants affected / at risk) | 43/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir Dipivoxil (N=80)
Acute pancreatitis (Gastrointestinal disorders) | 1
Nasal bone fracture (Musculoskeletal and connective tissue disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir Dipivoxil (N=80)
Retinopathy diabetic (Endocrine disorders) | 1
Xerophthalmia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Epigastric hunger pain (Gastrointestinal disorders) | 1
Epigastric pain (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Mouth dry (Gastrointestinal disorders) | 1
Oral submucous fibrosis (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Umbrical cord area pain (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Weakness generalized (General disorders) | 1
Liver fatty (Hepatobiliary disorders) | 1
Ascites (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Broncitis aggravated (Infections and infestations) | 1
Bronchitis chronic (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Alpha-fetoprotein increased (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 7
Creatine phosphokinase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Finger sprain (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Musculoskeletal and connective tissue disorders) | 1
Left wrist pain (Musculoskeletal and connective tissue disorders) | 1
Left knee pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain neck/shoulder (Musculoskeletal and connective tissue disorders) | 1
Right middle finger pain (Musculoskeletal and connective tissue disorders) | 1
Epidermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Numbness (Nervous system disorders) | 1
Tingling skin (Nervous system disorders) | 1
Vertigo (Nervous system disorders) | 1
Common cold (Respiratory, thoracic and mediastinal disorders) | 4
Coughing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.